CLINICAL TRIAL: NCT06758232
Title: Effects of a Neck Education Program in Parents of Children With Disabilities: A Single-Blind Randomized Controlled Trial
Brief Title: Neck Education for Parents of Disabled Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Dr. Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAEU-T.ATAHAN-008
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Chronic Neck Pain
Keywords: Chronic neck pain; Functional disability; Neck education; Parents of children with disabilities
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Study Group (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — It will consist of sessions that include neck anatomy, biomechanics, proper posture, ergonomics and neck exercise training.
  Arms: Study Group

SUMMARY:
Objective: Parents of children with disabilities are at risk of musculoskeletal pain, postural disorders, and functional limitations due to caregiving responsibilities and physical demands. This study aimed to evaluate the effects of a neck education program in parents of children with disabilities who have chronic neck pain.

Method: This single-blind randomized controlled trial included 62 parents diagnosed with chronic neck pain (intervention group: n=30; control group: n=32). The intervention group received a neck education program, while the control group did not receive any training. The program was implemented over five consecutive days and consisted of five 60-minute sessions. Neck pain intensity was assessed using the Visual Analog Scale (VAS) and the Short-Form McGill Pain Questionnaire (SF-MPQ); functional disability using the Neck Disability Index (NDI); spinal curvature using the Spinal Mouse device; posture using the Corbin Posture Assessment Scale (CPAS); physical activity level using the International Physical Activity Questionnaire-Short Form (IPAQ-SF); and quality of life using the SF-36. Assessments were conducted before and 12 weeks after the intervention. Data were analyzed using two-way mixed-design analysis of variance (ANOVA).

Results: At baseline, no significant differences were found between groups for any parameter (p > 0.05). After the intervention, the intervention group showed a significant improvement in NDI scores (p < 0.001), whereas no significant changes were observed in other parameters (p > 0.05).

Conclusion: The neck education program was found to be effective in reducing functional disability among parents of children with disabilities who experience chronic neck pain.

Keywords: Chronic neck pain; Functional disability; Neck education; Parents of children with disabilities

ELIGIBILITY:
Inclusion Criteria:

* Volunteer parents between the ages of 18-65, with spinal problems and chronic pain, pain lasting longer than 3 months, no inflammatory pain, no pain originating from abdominal-pelvic organs will be included in the study.

Exclusion Criteria:

* Individuals with acute fractures and malignancies, cervical disc herniation, those who have undergone surgical operations in the cervical region or spine, those with upper extremity pathologies, and those with rheumatological, neurological and psychological disorders will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Assessment of Neck Pain | 20 weeks
  Visual Analog Scale (VAS): VAS is a measurement generally used to assess pain intensity. VAS is a scale consisting of 10 cm horizontal lines numbered from 0 to 10. The "0" point indicates no pain; the "10" point indicates unbearable pain. The pain intensity felt by caregivers in their spine will be assessed with VAS. Participants will be asked to score the pain intensity felt during rest, activity and sleep between 0 and 10, and the results will be recorded.
Assessment of Neck Pain | 20 weeks
  Mc-Gill Melzack Pain Scale (MMAS): Participants' pain will be measured multidimensionally with MMAS. MMAS consists of 4 sections. The first section includes questions about the area of pain the patient has, the second section evaluates the pain in terms of perception and sensation, the third section includes questions about the relationship between pain and time, and the fourth section includes questions about the severity of pain. The scale is a 4-point Likert-type scale, and each item is scored between 0 and 3 (0: no pain; 3: the most severe pain), and a high total score indicates a high level of pain. The total pain score varies between 0 and 45 (0: no pain; 45: the most severe pain).
Neck Disability Assessment | 20 weeks
  The neck functionality of the participants will be assessed with the Neck Disability Index (NDI), which has validity and reliability. The index, which assesses daily living activities and symptoms, consists of a total of 10 sections. These sections include pain level, personal care, weight bearing, reading, headache, concentration, work life, driving, sleep status and recreational activities. A score between 0-4 is interpreted as no disability, a score between 5-14 is interpreted as mild disability, a score between 15-24 is interpreted as moderate disability, a score between 25-34 is interpreted as severe disability and a score above 35 is interpreted as total disability.
Evaluation of Spinal Curvature | 20 weeks
  Spinal Mouse (SM) is a computer-aided handheld electromechanical device. SM is a measurement tool developed to determine spinal column alignment, segmental and total curvatures, and vertebral motion angles in many planes. SM is a clinically applicable, valid, and objective method. In our study, the Idiag brand SM device will be used. The participants' clothes will be removed and measurements will be made with SM between the C7 (cervical) and S3 (sacral) regions. The data obtained from the measurement will be transferred to the computer via a wireless connection. On the computer, the data will be analyzed via the program and interpreted by the consultant.
Posture Evaluation | 20 weeks
  Posture analysis will be done with the CPAS (Corbin Posture Analysis Scale) prepared by Corbin and his friends. The participant will be evaluated with this scale in the posture analysis table from the lateral and posterior observations. The scale is scored between 0 and 3 (0: none; 3: severe) according to the severity of the disorder. The scores obtained by observing from the posterior and lateral are collected and classified in the final state (Poor ≥12; moderate 8-11; good 5-7; very good 3-4; excellent 0-2).
Physical Activity Evaluation | 20 weeks
  The physical activity level of the participants will be assessed with the International Physical Activity Questionnaire (IFQQ). The scale provides information about the time spent in sitting, walking, moderate and vigorous activities. The participants were asked how many days and how many minutes/hours they did vigorous and moderate exercise, walked and sat in the last 7 days. The criteria for evaluating the activities are based on the fact that each can be done for at least 10 minutes. A value called "MET minutes/week" is obtained by multiplying the minutes, days and metabolic equivalent (MET) values. The physical activity level is classified as physically inactive (<600 MET-min/week), low (minimally active) (600-3000 MET-min/week) and sufficient physical activity level for health (very active) (>3000 MET-min/week).
Assessment of Quality of Life | 20 weeks
  The Short Form-36 Quality of Life Scale (SF-36) will be used to assess quality of life. The scale consists of 8 different sub-dimensions (social function, physical function, emotional role difficulty, physical role difficulty, vitality (energy), pain, mental health, and general health) and a total of 36 items. Sub-groups are evaluated between 0-100 points, and "0 points" indicates poor health status, and "100 points" indicates good health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Atahan Turhan, Kırşehir, Merkez, Turkey (Türkiye)